CLINICAL TRIAL: NCT04311268
Title: Follow Fever to Decide: Determination of an Algorithm to Quantify and Qualify the Circadian Rhythmicity
Brief Title: Follow Fever to Decide
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Slb Pharma (Other)
Collaborators: Université de Caen Normandie (Other); Capital Innovation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: F2D
Record Dates: First submitted 2020-03-12; First posted 2020-03-17 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Body Temperature Changes
Keywords: Body Temperature; Circadian Rhythm
MeSH Terms: conditions — Body Temperature Changes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Observational (Experimental): Comparison of the core temperature obtained during 24-48 h with eCelsius and with F2D armband in different life situations.
  Interventions: Device: F2D armband

INTERVENTIONS:
Device: F2D armband — Comparison of the core temperature obtained during 24-48 h with eCelsius and with F2D armband in different life situations.

SUMMARY:
Body temperature is one of the markers of biological rhythms. The precise determination of the functioning of the biological clock for an individual is essential to understanding his physiological state at a given time. This condition is dependent on the "timing" of its central clock on the time scale (chronotype). The provision of a simple-to-use (F2D cuff), non-invasive and time-dependable temperature tool and the creation of appropriate algorithms would allow access to the operation of the central clock and open up many therapeutic applications.

DETAILED DESCRIPTION:
While the measurement of body temperature is one of the first self-diagnosis gestures at home, it is unanimously agreed by healthcare professionals that the measurement of non-invasive body temperature performed both in a hospital setting, in the office, that at home is very imprecise, or even false. As a result, temperature is only an indicator and is of little interest. Only the rectal thermometer and the telemetric capsule (e-CELSIUS® capsule to be ingested that allows a reliable and continuous measurement of gastrointestinal temperature without the intervention of the caregiver) are reliable tools, but they remain invasive and do not always allow for fully reliable follow-up over time. We propose to develop an algorithm integrated in an external, non-invasive cuff, allowing the continuous recording of body temperature.

In addition, body temperature is one of the markers of biological rhythms. The precise determination of the functioning of the biological clock for an individual is essential to understanding his physiological state at a given time. This condition is dependent on the "timing" of its central clock on the time scale (chronotype). The provision of a simple-to-use (F2D cuff), non-invasive and time-dependable temperature tool and the creation of appropriate algorithms would allow access to the operation of the central clock and open up many therapeutic applications.

This work proposes to validate the tool on the one hand and on the other to use this tool to produce the elements necessary for monitoring the functioning of the central biological clock.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female,
* Between 18 and 40 years of age for the WP I and II phases, and between 18 and 80 years of age for the WP III phase,
* Having an BMI within the range [18.5; 24.9] kg/m² for the Work Package I and II phases, and between [18.5; 34.9] kg/m² for the Work Package III phase,
* Beneficiary of the social security,
* Provided informed consent for participation in the study.

Exclusion Criteria:

* Presenting an acute pathology,
* Chronic pathology not followed and balanced,
* Having intestinal disorders (diverticles, disorders of the motility of the digestive tract, ...) or having undergone surgery at the gastrointestinal level,
* With known swallowing disorders,
* Having an alcohol dependence (more than 28 alcohol units per week), benzodiazepines or any illicit product,
* Smoking more than 5 cigarettes per day,
* Working nights or shift work,
* Simultaneous participation in other clinical research or participation in another clinical study for which the exclusion period has not ended.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2020-03-13 (Actual); Primary Completion 2021-12-18 (Actual); Study Completion 2021-12-18 (Actual)

PRIMARY OUTCOMES:
WP1 (body temperature) | 24 hours
  Comparison of the body temperature obtained by the e-CELSIUS® system with the body temperature obtained with the F2D system in 2 situations : during an exercice, to rise the core temperature, and during a nap taken in the afternoon to reduce it.
WP2 (body temperature) | 48 hours
  To continuously record the internal and external body temperature obtained with the e-CELSIUS® system and the F2D cuff for 48 hours to obtain a corpus of data allowing algorithm productions being able to quantify and qualify the circadian rhythmicity and determine the chronotype of normo-weighted subjects.
WP3 (body temperature) | 48 hours
  To continuously record the internal and external body temperature obtained with the e-CELSIUS® system and the F2D cuff for 48 hours to obtain a corpus of data allowing algorithm productions being able to quantify and qualify the circadian rhythmicity and determine the chronotype of subjects with varying ages and body sizes .

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratoire COMETE UMR-S 1075, Caen, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mazerolle SM, Ganio MS, Casa DJ, Vingren J, Klau J. Is oral temperature an accurate measurement of deep body temperature? A systematic review. J Athl Train. 2011 Sep-Oct;46(5):566-73. doi: 10.4085/1062-6050-46.5.566. PMID 22488144
- [Background] Weed HG. Review: Peripheral thermometers do not have clinically acceptable accuracy for measuring core body temperature. Ann Intern Med. 2016 Mar 15;164(6):JC32. doi: 10.7326/ACPJC-2016-164-6-032. No abstract available. PMID 26974732